CLINICAL TRIAL: NCT02409485
Title: Improving Self-Management in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hoda Badr, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 12-1641; R21CA178478 (NIH); H-48778 (Other: Baylor College of Medicine)
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Head and Neck Cancer
Keywords: self-management; head and neck cancer; psychosocial intervention; couples
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Couples Skill-Training (CST) (Experimental): CST provides education about acute and long-term side-effects of HNC and teaches: 1) self-management skills to control/prevent side-effects; 2) communication skills to facilitate coordination of care; and, 3) strategies to improve communal coping and confidence in the ability to work as a team.
  Interventions: Behavioral: Couples Skill-Training (CST)
- Usual Medical Care (UMC) (No Intervention): Patients receive standard symptom management education by their health care team.

INTERVENTIONS:
Behavioral: Couples Skill-Training (CST) — Patients and partners each receive a workbook and 6 one-hour telephone sessions with a Masters level trained interventionist. Manual content is tailored based on role (patient or partner). Couples participate together via speaker phone for half the sessions and patients and partners receive separate (individual) intervention calls for the other half of the sessions.
  Arms: Couples Skill-Training (CST)

SUMMARY:
By teaching skills to improve the coordination of care and support in couples coping with head and neck cancer (HNC), this couple-based psychosocial intervention holds great promise for improving self-management, reducing costly hospitalizations and treatment interruptions, and improving both partners' quality of life. Home-based delivery will enhance future dissemination and outreach to those who do not have access to psychosocial services or live far away from their care centers. If found effective, the intervention may also have salutary downstream effects on the health and well-being of HNC patients and their partners.

DETAILED DESCRIPTION:
Patients treated with radiation (XRT) for head and neck cancers (HNCs) experience significant side effects such as abnormally reduced salivation, difficulty swallowing, and taste changes even after they have been definitively treated. To control side effects and minimize discomfort, intensive self-care protocols are prescribed, but adherence is poor. Partners (spouses/significant others) can play a critical role in supporting adherence, but often lack knowledge, experience high rates of distress, and display poor communication (e.g., critical or controlling), that can interfere with patient self-care. The investigators have developed a home-based couples skills-training (CST) intervention that teaches: 1) self-management skills to control/prevent side-effects; 2) communication skills to facilitate coordination of care and support; and 3) strategies to improve communal coping and confidence in the ability to work as a team. The goal is to reduce healthcare utilization and improve multiple domains of patient and partner QOL. Specific aims are to: develop and evaluate the content and materials of the CST intervention (AIM 1) and evaluate its feasibility and acceptability (AIM 2). The multidisciplinary team will review and evaluate the content we have already developed based on the ongoing work with HNC couples (K07). Once content is finalized, tailored manuals will be developed for patients and partners and evaluated through two focus groups (AIM 1). The investigators expect that most couples (> 60%) approached will agree to participate and that CST will be well-accepted (AIM 2). Knowledge gained will be used to refine CST and to collect data on effect sizes and variation for a larger trial. Innovation: CST takes a multiple-behavioral approach to addressing and preventing HNC treatment side effects and, in the process, seeks to improve multiple domains of QOL. It is also the first program in HNC that actively involves both members of the couple to address barriers in the home environment in which self-management occurs. Finally, this study conceptualizes the couple relationship as a resource and leverages that resource to improve patient care and outcomes. Impact: Home-based delivery will enhance future dissemination and outreach to the target population. Overall, CST holds great promise for improving patient self-management behaviors, reducing costly hospitalizations and treatment interruptions, and improving multiple aspects of patient and partner QOL.

ELIGIBILITY:
Inclusion Criteria:

* patient is initiating radiotherapy for HNC
* patient has Karnofsky score > 50 (ambulatory & capable of self-care)
* patient lives with a partner (spouse/significant other - includes homo- and heterosexual couples)
* patient/partner is able to provide informed consent
* patient/partner is > age 18.

Exclusion Criteria:

* patient has significant comorbidities (e.g., HIV, transplant), or another illness that may require hospitalization
* patient/partner cannot read or communicate using spoken English.
* individuals with diminished mental capacity
* prisoners
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of the CST intervention as assessed by recruitment and retention rates | 6 months
  recruitment and retention rates
Acceptability of the CST intervention as assessed by the program evaluation questionnaire | 6 months
  satisfaction with the intervention by completing a program evaluation questionnaire developed by the study team that asks about perceived skills mastery and satisfaction with program content and logistics

SECONDARY OUTCOMES:
PROMIS short form anxiety and depression | 6 months
  measures distress with Patient Reported Outcomes Measurement Information System (PROMIS) short form for anxiety and depression
Patient QOL measured by MD Anderson Symptom Inventory - Head and Neck (MDASI-HN) | 6 months
  measures QOL for patients
Partners QOL measured by Short Form 12 (SF12) | 6 months
  measures QOL for partners
Short Form Dyadic Adjustment Scale (DAS7) | 6 months
  measures Relationship functioning
Healthcare utilization as assessed by number of hospitalizations and unplanned clinic visits | 6 months
  number of hospitalizations and unplanned clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Badr, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States